CLINICAL TRIAL: NCT05681676
Title: Is the Melanocortin System Involved in Inflammatory Resolution
Brief Title: Melanocortin Gene Expression in Lymphocytes of Polymyalgia Patients
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Michael Kruse Meyer, PhD, Aalborg University
Other Study IDs: N-20120074
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blod samples including lymphocytes and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood samples before and after standard of care of polymyalgia rheumatica — Blood samples were taken before glucocorticoid treatment and three months after.

SUMMARY:
Polymyalgia rheumatica (PMR) is a systemic inflammatory disorder with unknown etiology and overlapping symptoms with giant cell arthritis and rheumatoid arthritis (RA). The proteomic profile of PMR patients remains uncharacterized and biomarker studies very limited. The primary aim of this study was to thoroughly investigate the lymphocyte expression of melanocortin receptors, and the serum proteome during glucocorticoid treatment of PMR with a focus on acute-phase reactions, the complement system, and pro-inflammatory cytokines.

DETAILED DESCRIPTION:
Polymyalgia rheumatica (PMR) is a prototypic systemic inflammatory disease with overlapping symptoms similar to late onset rheumatoid arthritis (RA), giant cell arthritis (GCA), and cancer [1]. The etiology of PMR remains largely unknown, but it has been suggested that an age-related decline in the adaptive immune system might play a role in an over-compensatory inflammatory innate immune response [2]. Some genes and polymorphisms involved in initiation and regulation of inflammation have been associated with PMR [3,4] and polymorphisms are more predominant in the Northern European than Mediterranean population [5]. PMR has been somewhat successfully treated with glucocorticoids (e.g. prednisone) for more than half a century [6]. Due to the lack of causative molecular knowledge about the driving factors of inflammatory activation, and lack of treatment alternatives, glucocorticoids are still applied as the first line treatment today [7]. Relapses are common during standard glucocorticoid treatment [8], and randomized trials have failed to provide new treatment options [9,10]. However, recent progress in GCA treatment [11] have paved the way for biological treatment of PMR.

Only few serological biomarkers have been associated to PMR pathogenesis and disease activity while the pathogenesis of RA has been more thoroughly investigated. Hence, there is an unmet need to elucidate the pathophysiology of PMR. In this pilot-study, we therefore explored the potential to identify new serological markers at disease onset, which could be responsive to glucocorticoid treatment, which could be linked to PMR pathology. We did this using state-of-the-art quantitative proteomics profiling to investigate serum proteins from PMR patients before and after treatment with glucocorticoids for three months. In addition, we compared these patients with DMARD naïve RA patients, and healthy controls for potential molecular similarities. Hence, we applied advanced, qPCR to investigate lymphocyte expression, and mass spectrometry (MS) to measure serum proteins, and compared the results with serum cytokines.

ELIGIBILITY:
Inclusion Criteria:

* The PMR diagnosis fulfilled the ACR 1987 criteria [20]. Additional inclusion criteria were elevated CRP, and sedimentation rate, ultrasound verified synovitis [21], and ].

Exclusion Criteria:

* no cancer related findings on computed tomography (CT) of the abdomen, and chest X-ray to increase specificity as described by ACR 2012 classification criteria [22

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria ensured that the PMR patients had a high disease activity. After three months, the patients had obtained significant effect of the glucocorticoid treatment evaluated by physical examinations and clinical biochemistry values (Table 1).
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Melanocortin receptor expression | 3 months.
  Melanocortin receptor expression determined like previously: https://pubmed.ncbi.nlm.nih.gov/27434862/
Serum proteome | 3 months.
  Mass spectrometry investigated serum proteome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crowson CS, Matteson EL, Myasoedova E, Michet CJ, Ernste FC, Warrington KJ, Davis JM 3rd, Hunder GG, Therneau TM, Gabriel SE. The lifetime risk of adult-onset rheumatoid arthritis and other inflammatory autoimmune rheumatic diseases. Arthritis Rheum. 2011 Mar;63(3):633-9. doi: 10.1002/art.30155. PMID 21360492
- [Background] Pacheco MJ, Amado JA, Lopez-Hoyos M, Blanco R, Garcia-Unzueta MT, Rodriguez-Valverde V, Martinez-Taboada VM. Hypothalamic-pituitary-adrenocortical axis function in patients with polymyalgia rheumatica and giant cell arteritis. Semin Arthritis Rheum. 2003 Feb;32(4):266-72. doi: 10.1053/sarh.2003.49993. PMID 12621591
- [Background] Liang GC, Simkin PA, Hunder GG, Wilske KR, Healey LA. Familial aggregation of polymyalgia rheumatica and giant cell arteritis. Arthritis Rheum. 1974 Jan-Feb;17(1):19-24. doi: 10.1002/art.1780170105. No abstract available. PMID 4810661
- [Background] Owen CE, Buchanan RR, Hoi A. Recent advances in polymyalgia rheumatica. Intern Med J. 2015 Nov;45(11):1102-8. doi: 10.1111/imj.12823. PMID 26036315
- [Background] Salvarani C, Pipitone N, Versari A, Hunder GG. Clinical features of polymyalgia rheumatica and giant cell arteritis. Nat Rev Rheumatol. 2012 Sep;8(9):509-21. doi: 10.1038/nrrheum.2012.97. Epub 2012 Jul 24. PMID 22825731
- [Background] Behn AR, Perera T, Myles AB. Polymyalgia rheumatica and corticosteroids: how much for how long? Ann Rheum Dis. 1983 Aug;42(4):374-8. doi: 10.1136/ard.42.4.374. PMID 6882032
- [Background] Dejaco C, Singh YP, Perel P, Hutchings A, Camellino D, Mackie S, Abril A, Bachta A, Balint P, Barraclough K, Bianconi L, Buttgereit F, Carsons S, Ching D, Cid M, Cimmino M, Diamantopoulos A, Docken W, Duftner C, Fashanu B, Gilbert K, Hildreth P, Hollywood J, Jayne D, Lima M, Maharaj A, Mallen C, Martinez-Taboada V, Maz M, Merry S, Miller J, Mori S, Neill L, Nordborg E, Nott J, Padbury H, Pease C, Salvarani C, Schirmer M, Schmidt W, Spiera R, Tronnier D, Wagner A, Whitlock M, Matteson EL, Dasgupta B; European League Against Rheumatism; American College of Rheumatology. 2015 Recommendations for the management of polymyalgia rheumatica: a European League Against Rheumatism/American College of Rheumatology collaborative initiative. Ann Rheum Dis. 2015 Oct;74(10):1799-807. doi: 10.1136/annrheumdis-2015-207492. PMID 26359488
- [Background] Salvarani C, Cantini F, Niccoli L, Macchioni P, Consonni D, Bajocchi G, Vinceti M, Catanoso MG, Pulsatelli L, Meliconi R, Boiardi L. Acute-phase reactants and the risk of relapse/recurrence in polymyalgia rheumatica: a prospective followup study. Arthritis Rheum. 2005 Feb 15;53(1):33-8. doi: 10.1002/art.20901. PMID 15696567
- [Background] Salvarani C, Macchioni P, Manzini C, Paolazzi G, Trotta A, Manganelli P, Cimmino M, Gerli R, Catanoso MG, Boiardi L, Cantini F, Klersy C, Hunder GG. Infliximab plus prednisone or placebo plus prednisone for the initial treatment of polymyalgia rheumatica: a randomized trial. Ann Intern Med. 2007 May 1;146(9):631-9. doi: 10.7326/0003-4819-146-9-200705010-00005. PMID 17470831
- [Background] Kreiner F, Galbo H. Effect of etanercept in polymyalgia rheumatica: a randomized controlled trial. Arthritis Res Ther. 2010;12(5):R176. doi: 10.1186/ar3140. Epub 2010 Sep 20. PMID 20854662
- [Background] Stone JH, Tuckwell K, Dimonaco S, Klearman M, Aringer M, Blockmans D, Brouwer E, Cid MC, Dasgupta B, Rech J, Salvarani C, Schett G, Schulze-Koops H, Spiera R, Unizony SH, Collinson N. Trial of Tocilizumab in Giant-Cell Arteritis. N Engl J Med. 2017 Jul 27;377(4):317-328. doi: 10.1056/NEJMoa1613849. PMID 28745999
- [Background] Arnett FC, Edworthy SM, Bloch DA, McShane DJ, Fries JF, Cooper NS, Healey LA, Kaplan SR, Liang MH, Luthra HS, et al. The American Rheumatism Association 1987 revised criteria for the classification of rheumatoid arthritis. Arthritis Rheum. 1988 Mar;31(3):315-24. doi: 10.1002/art.1780310302. PMID 3358796
- [Background] Kermani TA, Warrington KJ. Advances and challenges in the diagnosis and treatment of polymyalgia rheumatica. Ther Adv Musculoskelet Dis. 2014 Feb;6(1):8-19. doi: 10.1177/1759720X13512450. PMID 24489611